CLINICAL TRIAL: NCT05942144
Title: Exercise-snacks: an Effective Strategy to Break Sitting Time and Improve Cardiometbaolic Health in Sedentary Overweight Office Workers
Brief Title: Exercise-snacks at Work: Impact on Cardiometabolic Parameters
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Post hoc power analysis results on the primary hypothesis during the preliminary analyses
Sponsor: University of Avignon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AU-062023-AVJ
Record Dates: First submitted 2023-06-19; First posted 2023-07-12 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Sedentary Time; Overweight and Obesity; Work-Related Condition
Keywords: brief intense exercise; vascular function; cardiorespiratory fitness
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise-snacks group (Experimental): They will perform a "exercise-snacks" program and receive information about physical activity
  Interventions: Other: Exercise-snacks program
- Control group (No Intervention): They will maintain their usual lifestyle until the end of the study

INTERVENTIONS:
Other: Exercise-snacks program — Subjects in the exercise-snacks group will perform 4 "exercise-snacks" sessions per working day for 4 weeks. These sessions will consist of 80 one-to-one walks to be completed as quickly as possible. They will also receive information about their attitudes to physical activity.
  Arms: Exercise-snacks group

SUMMARY:
The main objective is to measure the effects of intense brief exercise program in the workplace of administrative staff on the cardio-metabolic health

DETAILED DESCRIPTION:
Backgrounds: Very short (< 1 minute) and intense exercises, entitled "exercise-snacks", have been reported to be effective 1) in improving physical fitness over 6 weeks and 2) in improving vascular function and lowering blood glucose levels over one day. These studies were all carried out in the laboratory. The question therefore arises as to whether these acute vascular and metabolic benefits, as well as those on physical fitness, are sustainable over time following a chronic "exercise-snacks" program applicable in the professional environment to sedentary, overweight people.

Aims of this project is therefore to measure the effects of an "exercise-snacks" type physical activity program in the workplace of administrative staff on the cardio-metabolic health and sedentary behaviour of staff.

ELIGIBILITY:
Inclusion Criteria:

* administrative staff,
* age between 30 and 60,
* body mass index ≥25kg/m²,
* sedentary time ≥7h/day,
* minimum 3 working days on site,
* no known cardiovascular or metabolic pathology, social security affiliation or benefit,
* ability and willingness to give free, written and informed consent.

Exclusion Criteria:

* pregnant or breast-feeding women,
* anti-hypertensive treatment, beta-blockers and anti-diabetics,
* known contraindications to physical activity (articular, cardiac or other),
* exercise-induced asthma,
* lack of motivation of subjects posing problems of compliance and adherence to the exercise program,
* participation in a study in the preceding 3 months, ongoing participation in a clinical trial.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Changes in aerobic fitness | at inclusion, at the end of the 4-weeks program and 1 month following the end of the program
  Aerobic fitness will be assessed via the Chester step test's prediction of VO2max

SECONDARY OUTCOMES:
Adherence of staff in the experimental group by analyzing accelerometric data. | during the 4-weeks program
  Total number of exercise-snacks performed during the 4-week program by analysing accelerometers data
Intensity of exercise-snacks | during the 4-weeks program
  Heart rate during exercise-snacks in % heart rate max
Changes in flow mediated dilation of superficial femoral artery | at inclusion, at the end of the 4-weeks program
  measured by echocardiography (Vivid Q, GE) , in %
Changes in peak shear rate of superficial femoral artery | at inclusion, at the end of the 4-weeks program
  measured by echocardiography (Vivid Q, GE) during hyperemia, in s-1
Changes in nitrate mediated dilation of superficial femoral artery | at inclusion, at the end of the 4-weeks program
  by echocardiography (Vivid Q, GE), in %
Changes in superficial femoral artery compliance | at inclusion, at the end of the 4-weeks program
  by echocardiography (Vivid Q, GE), in mm2 mmHg-1
Changes in carotid intima-thickness | at inclusion, at the end of the 4-weeks program
  by echocardiography (Vivid Q) in mm
Changes in carotid compliance | at inclusion, at the end of the 4-weeks program
  by echocardiography (Vivid Q) in mm2 mmHg-1
Changes in carotid-femoral pulse wave velocity | at inclusion, at the end of the 4-weeks program
  by Sphygmocor, in m.s-1
Changes in post-occlusive skin perfusion | at inclusion, at the end of the 4-weeks program
  by Laser Doppler (Perimed), in perfusion unit, in area under the curve, in time to peak
Changes in blood pressure | at inclusion, at the end of the 4-weeks program and 1 month following the end of the program
  systolic, diastolic, mean and pulsed
Changes in mean amplitude of glycemic excursions | one week before the beginning of the program and the first week of the program and the 2 lastest weeks of the program
  measured by continuous glucose monitoring (FreeStyle), in mmol.L-1
Changes in heart rate | between the beginning and end of the 4-week exercise program and 4 weeks after the program.
  Heart rate at rest, at the end of the Chester step test and during exercise
Changes in level of habitual physical activity | between the start and end of the 4-week exercise program and 4 weeks after the program
  Physical Activity questionnaire
Changes in fat mass | between the start and end of the 4-week exercise program and 4 weeks after the program
  measured by InBody, in kg
Changes in lean mass | between the start and end of the 4-week exercise program and 4 weeks after the program
  measured by InBody, in kg
Change in physical activity behaviour at work of staff | between the start and end of the 4-week exercise program.
  Theory of planned behavior questionnaire, score range from 20 to 80 with higher scores mean a better outcome.
Changes in rating of perceived exertion | between the start and end of the 4-week exercise program and 4 weeks after the program
  measured during the Chester test, score range from 7 to 20 with higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Agnès VINET, Principal Investigator — Avignon University - LaPEC
Locations (1):
- Avignon University, Avignon, France